CLINICAL TRIAL: NCT04837573
Title: Evaluating the Feasibility and Acceptability of a Therapeutically-Grounded Virtual Sister Circle Intervention for Black Women With Depressive Symptoms
Brief Title: Feasibility & Acceptability of a Virtual Sister Circle Intervention for Black Women With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kia Skrine Jeffers, PhD, RN, PHN (Other)
Responsible Party: Sponsor-Investigator, Kia Skrine Jeffers, PhD, RN, PHN, Assistant Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-002949
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Depressive Symptoms; Depression
Keywords: Sister Circle; Black Women
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Intervention, Weeks 1-8 (Experimental): During Weeks 1-8, Group 1 receives the Intervention and Group 2 receives no treatment.
  Interventions: Behavioral: Sister Circle protocol
- Group 2 Intervention, Weeks 9-16 (Active Comparator): During Weeks 9-16, Group 2 receives the Intervention and Group 1 receives no treatment.
  Interventions: Behavioral: Sister Circle protocol

INTERVENTIONS:
Behavioral: Sister Circle protocol — The intervention is an 8-week, therapeutically-informed protocol.

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of a protocol for middle- and older-aged Black women with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black or African American
* Identify as female
* Age 40 years and older
* Community-dwelling
* Self-report of experiencing depressive symptoms
* Ability to commit to the 8-week intervention
* Access to Zoom
* Speak and read English

Exclusion Criteria:

* Have a diagnosis of bipolar, but is not taking medication for the condition
* Experiencing psychosis

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females
Enrollment: 30 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Recruitment, completion, and retention rates of participants | 16 weeks
  80 percent recruitment, 80 percent completion, and 75 percent retention
Assess Acceptability according to the Theoretical Framework of Acceptability | 16 weeks
  Qualitative assessment of Acceptability. The interview guide will be organized according to the constructs of the Theoretical Framework of Acceptability. Methodological conventions of qualitative description will be used to analyze the data.

SECONDARY OUTCOMES:
Changes in Perceived Stress Scale (PSS) from baseline at 8 weeks and 16 weeks | baseline, 8 weeks, 16 weeks
  Exploratory description of effect sizes
Changes in Positive and Negative Affect Schedule (PANAS) Scale from baseline at 8 weeks and 16 weeks | baseline, 8 weeks, 16 weeks
  Exploratory description of effect sizes
Changes in Acceptance and Action Questionnaire II (AAQ-II) from baseline at 8 weeks and 16 weeks | baseline, 8 weeks, 16 weeks
  Exploratory description of effect sizes

CONTACTS AND LOCATIONS:
Overall Officials: Kia Skrine Jeffers, PhD, RN, PHN, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States